CLINICAL TRIAL: NCT01099423
Title: Randomized Phase III Trial Comparing Immediate Versus Deferred Nephrectomy in Patients With Synchronous Metastatic Renal Cell Carcinoma
Brief Title: Immediate Surgery or Surgery After Sunitinib Malate in Treating Patients With Metastatic Kidney Cancer
Acronym: SURTIME
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Wales Cancer Trials Unit (Other); Canadian Urologic Oncology Group (Other); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-30073; EU-21022; PFIZER-EORTC-30073
Record Dates: First submitted 2010-04-06; First posted 2010-04-07 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Kidney Cancer
Keywords: clear cell renal cell carcinoma; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Gene Expression Profiling

ARMS (2):
- Immediate nephrectomy (Active Comparator): Surgery followed by Sunitinib
  Interventions: Genetic: gene expression analysis; Other: biologic sample preservation procedure; Other: laboratory biomarker analysis; Procedure: therapeutic conventional surgery
- Deferred nephrectomy (Experimental): Sunitinib (3 cycles) followed by surgery followed by Sunitinib
  Interventions: Procedure: timing of surgery; Genetic: gene expression analysis; Other: biologic sample preservation procedure; Other: laboratory biomarker analysis

INTERVENTIONS:
Procedure: timing of surgery
  Arms: Deferred nephrectomy
Genetic: gene expression analysis
Other: biologic sample preservation procedure
Other: laboratory biomarker analysis
Procedure: therapeutic conventional surgery
  Arms: Immediate nephrectomy

SUMMARY:
RATIONALE: Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving sunitinib malate before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving sunitinib malate after surgery may kill any tumor cells that remain after surgery. It is not yet known whether undergoing immediate surgery or surgery after sunitinib malate is more effective in treating patients with metastatic kidney cancer.

PURPOSE: This randomized phase III trial is studying immediate surgery to see how well it works compared with surgery after sunitinib malate in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if immediate versus deferred nephrectomy has an effect on disease control in patients with resectable, synchronous, metastatic renal cell carcinoma treated with sunitinib malate.
* To identify potential response criteria based on histopathology and molecular research on tumor tissue.

OUTLINE: This is a multicenter study. Patients are stratified according to WHO performance status (0 vs 1), number of metastatic sites (1 vs 2 or more), and institution. Patients are randomized to 1 of 2 treatment arms.

* Arm I (immediate nephrectomy): Patients undergo cytoreductive nephrectomy. Beginning 4 weeks after surgery, patients receive oral sunitinib malate once daily on days 1-28. Treatment with sunitinib malate repeats every 6 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (deferred nephrectomy): Patients receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 6 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. About 1 day after completion of sunitinib malate, patients undergo cytoreductive nephrectomy. Patients then receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

Some patients undergo tumor tissue collection at baseline and at time of surgery to assess possible differences in gene expression. Patients also undergo blood sample collection periodically to evaluate the potential impact of serum proteins on the clinical outcome. Samples are then stored for future studies.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell cancer (RCC)

  * Clear-cell subtype with a resectable asymptomatic in situ primary

    * Asymptomatic primary is defined as the absence of symptoms* which can be exclusively assigned to the primary tumor such as flank pain and/or gross hematuria necessitating blood transfusion NOTE: *Para-neoplastic symptoms cannot be assigned to the primary tumor alone in metastatic disease, they are not included in this definition.
    * No symptomatic primary tumor necessitating nephrectomy
* Resectable primary tumor

  * Bulky locoregional lymph node metastases larger than the primary tumor allowed provided resectability of the lymph nodes is surgically feasible
* Metastatic RCC

  * Distant metastases are not completely resectable at the time of surgery or during an additional intervention
  * No multiple distant lesions at one site
  * No bone-only metastases
* Measurable disease, both primary and metastatic, according to RECIST 1.1 criteria
* Planning to receive sunitinib malate as background therapy
* Patients with > 3 of the following surgical risk factors are not eligible:

  * Serum albumin CTCAE v 4.0 grade 2 or worse
  * Serum LDH > 1.5 times upper limit of normal
  * Liver metastases
  * Symptoms at presentation due to metastases
  * Retroperitoneal lymph node involvement
  * Supra-diaphragmatic lymph node involvement
  * Clinical stage T3 or T4 disease
* No clinical signs of CNS involvement

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* WHO performance status 0-1
* Life expectancy > 3 months
* WBC > 3.0 x 10^9/L
* Platelet count > 100 x 10^9/L
* Hemoglobin > 10.0 g/dL
* PT/PTT or INR ≤ 1.2 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* ALT ≤ 2.5 times ULN (≤ 5 times ULN if liver lesions)
* Serum calcium < 10.0 mg/dL
* Calculated or measured creatinine clearance > 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception 2 weeks before and during study treatment
* LVEF normal by MUGA scan or ECHO
* 12-lead ECG normal
* No serious cardiac illness (myocardial infarction and/or treatable or untreatable angina pectoris not responding to treatment) within the past 12 months
* No uncontrolled, high BP (≥ 150/100 mm Hg) despite optimal medical therapy
* No current pulmonary disease
* No active or uncontrolled infections, serious illnesses, malabsorption syndrome, or medical conditions, including patients with a history of chronic alcohol abuse, hepatitis, HIV, and/or cirrhosis
* No malignancies within the past 5 years except renal cell carcinoma, basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, resected incidental prostate cancer staged pT2 with Gleason Score ≤ 6 and postoperative PSA < 0.5 ng/mL, or patients with any history of malignancies who are disease-free for more than 5 years
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

PRIOR CONCURRENT THERAPY:

* Prior local radiotherapy for bone lesions allowed
* No prior systemic therapy for metastatic RCC
* No prior partial or total nephrectomy
* No concurrent systemic corticosteroid and/or other immunosuppressive systemic therapies
* No concurrent radiotherapy, except palliative radiotherapy
* No concurrent participation in another clinical trial testing treatments for any disease including renal cell carcinoma
* No other concurrent investigational or systemic therapy for metastatic RCC

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Overall progression-free survival

SECONDARY OUTCOMES:
Overall survival
Morbidity
Overall response to treatment in the deferred nephrectomy arm including the proportion of patients who become unresectable
Effect of nephrectomy on early progression in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Axel Bex, Study Chair — The Netherlands Cancer Institute; John B.A.G. Haanen, Study Chair — The Netherlands Cancer Institute
Locations (29):
- Belgium (7):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Cliniques Universitaires St. Luc, Brussels
  - Hôpitaux Universitaires Bordet-Erasme - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Virga Jesse Hospital, Hasselt
  - AZ Groeninghe - Campus Loofstraat, Kortrijk
  - AZ Damiaan - Campus Sint-Jozef, Ostend
- Canada (6):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - CHUM - Pavillon Saint-Luc, Montreal, Quebec
  - Montreal General Hospital, Montreal
  - The Ottawa Hospital, The Integrated Cancer Program- General Campus, Ottawa
  - University Health Network - Oci / Princess Margaret Hospital, Toronto
  - Diamond Health Care Centre, Vancouver
- San Camillo Forlanini Hospitals, Roma, Italy
- Netherlands (8):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Academisch Medisch Centrum - Universiteit van Amsterdam, Amsterdam
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - University Medical Center Groningen, Groningen
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Universitair Medisch Centrum - Academisch Ziekenhuis, Utrecht
- United Kingdom (7):
  - Royal United Hospital, Bath
  - University Hospitals Bristol NHS Foundation Trust - Bristol Haematology And Oncology Centre, Bristol
  - St. James'S University Hospital, Leeds
  - Barts and The London NHS Trust - St. Bartholomew'S Hospital, London
  - Imperial College Healthcare NHS Trust - Charing Cross Hospital, London
  - Christie NHS Foundation Trust, Manchester
  - Singelton Hospital, Swansea

REFERENCES:
- [Derived] Bex A, Mulders P, Jewett M, Wagstaff J, van Thienen JV, Blank CU, van Velthoven R, Del Pilar Laguna M, Wood L, van Melick HHE, Aarts MJ, Lattouf JB, Powles T, de Jong Md PhD IJ, Rottey S, Tombal B, Marreaud S, Collette S, Collette L, Haanen J. Comparison of Immediate vs Deferred Cytoreductive Nephrectomy in Patients With Synchronous Metastatic Renal Cell Carcinoma Receiving Sunitinib: The SURTIME Randomized Clinical Trial. JAMA Oncol. 2019 Feb 1;5(2):164-170. doi: 10.1001/jamaoncol.2018.5543. PMID 30543350
- [Derived] Leon L, Garcia-Figueiras R, Suarez C, Arjonilla A, Puente J, Vargas B, Mendez Vidal MJ, Sebastia C. Recommendations for the clinical and radiological evaluation of response to treatment in metastatic renal cell cancer. Target Oncol. 2014 Mar;9(1):9-24. doi: 10.1007/s11523-013-0304-7. Epub 2013 Dec 12. PMID 24338498
- [Derived] Winquist E, Rodrigues G. Open clinical uro-oncology trials in Canada. Can J Urol. 2012 Dec;19(6):6587-91. No abstract available. PMID 23228299